CLINICAL TRIAL: NCT04294251
Title: A Double-blind, Randomized, Placebo-controlled, Multi-center, Phase Ⅲ Study to Evaluate the Efficacy and Safety of NABOTA® in Subjects With Benign Masseteric Hypertrophy
Brief Title: Efficacy and Safety of DWP450 in Subjects With Benign Masseteric Hypertrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP450301
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2020-07

CONDITIONS: Benign Masseteric Hypertrophy
MeSH Terms: interventions — DWP450

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP450 (Experimental)
  Interventions: Drug: DWP450
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWP450 — Botulinum toxin type A(DWP450) will be administered intramuscularly to the bilateral masseter muscles on Day 1.
  Arms: DWP450
Drug: Placebo — Placebo(Normal Saline) will be administered intramuscularly to the bilateral masseter muscles on Day 1.
  Arms: Placebo

SUMMARY:
This Study is A Double-blind, Randomized, Placebo-controlled, Multi-center, Phase III Study to Evaluate the Efficacy and Safety of DWP450 in Subjects With Benign Masseteric Hypertrophy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject over 18 years of age and written informed consent is obtained.
2. Subject with Benign Masseter Hypertrophy.
3. Subject who has Bisymmetry of masseter at visual assessment.
4. Subjects who meets thickness of Masseter muscle by ultrasonography.
5. Subjects who can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. Diagnosis of Myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
2. Subject who got any facial aesthetic procedure (e.g. surgery, laser, thread treatment etc.) in lower facial area within 52 weeks prior to the study entry.
3. Subject who had previously received botulinum toxin within 12 weeks prior to the study entry.
4. Subject with known hypersensitivity to botulinum toxin.
5. Subject who are pregnant or lactating or found pregnancy though the urine or sebum test or disagreed to avoid pregnancy during study period.
6. Subjects who are not eligible for this study at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in masseter muscle thickness | 12 weeks
  Change from baseline in masseter muscle thickness by Ultrasonography

SECONDARY OUTCOMES:
Change from baseline in masseter muscle thickness | 24 weeks
  Change from baseline in masseter muscle thickness by Ultrasonography
Change from baseline in lower face volume | 24 weeks
  Change from baseline in lower face volume by 3D digital imaging
Overall satisfaction of subject: questionnaire | 24 weeks
  Subject satisfaction assessment using a scale ranging from very dissatisfied to very satisfied by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-ang University Hospital, Seoul, South Korea